CLINICAL TRIAL: NCT03606902
Title: Continuous Epidural Fentanyl Infusion Step-down Tapering Dose; Sole Intraoperative Analgesic Modality for Precious Single Kidney Patient.
Brief Title: Continuous Epidural Fentanyl- Low Dose Bupivacaine Infusion Analgesia for Precious Single Kidney Patient.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: R.18.01.4 - 20
Record Dates: First submitted 2018-07-07; First posted 2018-07-31 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-03

CONDITIONS: Postoperative Analgesia
Keywords: Epidural, Fentanyl, Kidney, Continuous, nephrotoxic.
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Intervention Model Description: double blinded randomized controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: • double blinded randomized controlled study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group f): (Active Comparator): Intervention:
  1. Procedure: Epidural catheter insertion
  2. Drug: Epidural 15 ml of 0.0625%bupivacaine with 1 µg /Kg Fentanyl ,then continuous epidural infusion of fixed volume 10 ml of 0.0625% bupivacaine +1 µg/Kg/h Fentanyl for the next 6 hours .
  Interventions: Procedure: Group f : Epidural catheter insertion; Drug: Group F: Continous epidural infusion of bupivacaine plus fentanyl
- (Group Lf): (Active Comparator): Intervention:
  1. Procedure:Epidural catheter insertion
  2. Drug: Epidural injection 15 ml of 0.0625%bupivacaine with 1 µg/Kg Fentanyl initial bolus, then 1st hour continuous IV infusion of 10ml of 0.0625%bupivacaine +1 µg/Kg/h Fentanyl ,2nd hour 10ml of 0.0625%bupivacaine + 0.5 µg/Kg/h Fentanyl , then next 4 hours10 ml of 0.0625%bupivacaine with + 0.25 µ g/Kg/h Fentanyl.
  Interventions: Drug: Group LF :Continous epidural infusion of decreasing doses of fentanyl plus pubivacaine; Procedure: Group L f : Epidural catheter insertion

INTERVENTIONS:
Procedure: Group f : Epidural catheter insertion — Infiltrate the skin with local anesthetic lidocaine approximately 1 cm lateral to the inferior aspect of the targeted spinous process , epidural needle tip is midline at the junction of the lamina and spinous process . The needle is withdrawn and advanced with the same medial angle but in small increments cephalad to the same depth. Either bone or ligamentum flavum is contacted. If bone is contacted, the needle is redirected cephalad and advanced. If bone is no longer contacted and the depth exceeds the depth previously noted, the epidural needle stilette is removed. loss-of-resistance syringe is attached to the needle Once attained, stabilize the epidural needle and thread the catheter. Secure the catheter using a sterile locking device and adherent dressings.
  Arms: (Group f):
Drug: Group F: Continous epidural infusion of bupivacaine plus fentanyl — Epidural injection of bolus of 15 ml total Volume of 0.0625%bupivacaine with 1 µg /Kg Fentanyl initial bolus, then from the 1st hour continuous epidural infusion of 0.0625% bupivacaine with µ/Kg/h Fentanyl fixed for the next 5 hour during operation and in the recovery room after recovery of general anesthesia then stop epidural infusion. (Total infusion time 6 hours=maximum hours needed for nephrectomy surgery)
  Arms: (Group f):
Drug: Group LF :Continous epidural infusion of decreasing doses of fentanyl plus pubivacaine — Epidural injection of bolus of 15 ml total Volume of 0.0625%bupivacaine with 1 µg/Kg Fentanyl initial bolus, then continuous IV infusion of 0.0625%bupivacaine with 1 µg/Kg/h Fentanyl for the 1st hour then continuous epidural infusion of 0.0625%bupivacaine with 0.5 µg/Kg/h Fentanyl during the 2nd hour, then 0.0625%bupivacaine with 0.25 µ g/Kg/h Fentanyl for the 3rd hour then continue the same infusion volume and dose (0.0625%bupivacaine with 0.25Mg/Kg/h Fentanyl) for the next 3 hours during operation and in the recovery room after recovery of general anesthesia then stop epidural infusion. (Total infusion time 6 hours=maximum hours needed for nephrectomy surgery)
  Arms: (Group Lf):
Procedure: Group L f : Epidural catheter insertion — Infiltrate the skin with local anesthetic lidocaine approximately 1 cm lateral to the inferior aspect of the targeted spinous process , epidural needle tip is midline at the junction of the lamina and spinous process . The needle is withdrawn and advanced with the same medial angle but in small increments cephalad to the same depth. Either bone or ligamentum flavum is contacted. If bone is contacted, the needle is redirected cephalad and advanced. If bone is no longer contacted and the depth exceeds the depth previously noted, the epidural needle stilette is removed. loss-of-resistance syringe is attached to the needle Once attained, stabilize the epidural needle and thread the catheter. Secure the catheter using a sterile locking device and adherent dressings.
  Arms: (Group Lf):

SUMMARY:
Open surgical nephrectomy is associated with sever postoperative pain mandating alternative strong ,renal safety, minimal side effects, and minimal rescue systemic analgesics , continuous Epidural Fentanyl infusion in a dose step down tapering manner would produce hemodynamic stability with effective analgesia in nephrectomy surgery without using nephrotoxic analgesic drugs such as NSAIDs .The study proposal: Continuous Epidural Fentanyl infusion in a dose step down tapering manner with the least analgesic LA dose is enough intraoperative non nephrotoxic analgesic modality with good intraoperative(IO) Hemodynamic stability & less postoperative complications in patients subjected to nephrectomy surgery with remaining single precious kidney. Aim of the work: Intraoperative analgesic technique avoiding polymodal analgesia that utilize the nephrotoxic NSAIDs, To have a NSAIDs free surgery by using a Continuous IO effective & safe lipophilic opioid analgesia especially in nephrectomy surgery that leaves the patient with a single precious healthy kidney that has to be well perfused and totally protected from any nephrotoxic drugs with rapid recovery and less PO complications

DETAILED DESCRIPTION:
• Introduction Open surgical nephrectomy is associated with sever postoperative pain mandating alternative strong ,renal safety, minimal side effects, and minimal rescue systemic analgesics , continuous Epidural Fentanyl infusion in a dose step down tapering manner would produce hemodynamic stability with effective analgesia in nephrectomy surgery without using nephrotoxic analgesic drugs such as NSAIDs .The study proposal: Continuous Epidural Fentanyl infusion in a dose step down tapering manner with the least analgesic LA dose is enough intraoperative non nephrotoxic analgesic modality with good intraoperative(IO) Hemodynamic stability & less postoperative complications in patients subjected to nephrectomy surgery with remaining single precious kidney. Aim of the work: Intraoperative analgesic technique avoiding polymodal analgesia that utilize the nephrotoxic NSAIDs, To have a NSAIDs free surgery by using a Continuous IO effective & safe lipophilic opioid analgesia especially in nephrectomy surgery that leaves the patient with a single precious healthy kidney that has to be well perfused and totally protected from any nephrotoxic drugs with rapid recovery and less PO complications. Material & Methods 50 adult patients, ASA I-III of both genders were randomly allocated into two groups each of 25 patients Control group (Group f):: using an epidural catheter technique with epidural catheter set, and at L1-2 insertion level directed up to cover up to T6 sensory level, Epidural injection of 15 ml total Volume of 0.0625%bupivacaine with 1µ/Kg/h Fentanyl for the 1st hour then 10ml of 0.0625% bupivacaine with 1µ/Kg/h Fentanyl for the next 5 hour then stop epidural infusion. Study group -Less Epidural Fentanyl group-(Group Lf): using an epidural catheter technique with epidural catheter set, and at L1-2 insertion level directed up to cover up to T6 sensory level, Epidural injection of 15 ml total Volume of 0.0625%bupivacaine with 1µ/Kg/h Fentanyl for the 1st hour then 10ml of 0.0625%bupivacaine with 0.5µ/Kg/h Fentanyl surgery then 3rd h 0.0625%bupivacaine with 0.25µ/Kg/h Fentanyl continue the same infusion volume and dose for the next 3 hours Preoperative preparation: After patient examination and consultation about any co-morbidities & explanation of the anesthetic procedures the consent will be taken after, clarification of VAS. Then 20 gage IV Catheter & Pre-loading by 500 ml Nacl0.9% solution over 30 minutes before anesthesia.

With the Patient in sitting position after skin disinfection and an 18-gauge epidural catheter was placed in the epidural space at T8-T9 or T9-T10 inter-space in both Groups of patients at T10-T11 or T11-T12 level, under local anesthesia, by an anesthesiology resident not involved in the study utilizing loss-of-resistance technique [9]. The study solutions were prepared by an anesthesiologist who was not involved in subsequent patient care or assessment. Using an epidural catheter set, to cover up to T6 sensory level, drug concentration 200 µ fentanyl (4ml)+ (5 ml) Bupivacaine 0.5% then add 31 ml sterile saline to have a total volume of 40 ml with concentration of 0.0625 with 5 µ fentanyl /ml of the cocktail solution. Then for every patient will calculate how much infusion will be based on body weight for example ( for a patient body weight 70kg ,1 µ/Kg/h infusion the volume will be 14 ml/h, 0.5 µ/Kg/h =7 ml/h,0.25 µ/kg/h =3.5 ml/h)

* Control group (Group f): Epidural injection of bolus of 15 ml total Volume of 0.0625%bupivacaine with 1µ/Kg Fentanyl initial bolus, then from the 1st hour continuous epidural infusion of 0.0625% bupivacaine with µ/Kg/h Fentanyl fixed for the next 5 hour during operation and in the recovery room after recovery of general anesthesia then stop epidural infusion.
* Study group -Less Epidural Fentanyl group-(Group Lf): Epidural injection of bolus of 15 ml total Volume of 0.0625%bupivacaine with 1 µg/Kg Fentanyl initial bolus, then continuous IV infusion of 0.0625%bupivacaine with 1 µg/Kg/h Fentanyl for the 1st hour then continuous epidural infusion of 0.0625%bupivacaine with 0.5 µg/Kg/h Fentanyl during the 2nd hour, then 0.0625%bupivacaine with 0.25 µ g/Kg/h Fentanyl for the 3rd hour then continue the same infusion volume and dose (0.0625%bupivacaine with 0.25µ/Kg/h Fentanyl) for the next 3 hours during operation and in the recovery room after recovery of general anesthesia then stop epidural infusion.
* Intraoperative management: After attaching basic monitoring NIBP cuff, Puls Oximeter probe, ECG, and EtCo2, Preoxygenation 5l O2 mask, for 5 minutes with the patient in sitting position with neck and upper back flexed. Widely prepare and drape the targeted thoracic segment(s) using sterile technique. Infiltrate the skin and subcutaneous tissues with local anesthetic approximately 1 cm lateral to the inferior aspect of the targeted spinous process with a 1.5- inch 25-gauge needle. With the infiltration needle, contact the ipsilateral lamina or transverse process and anesthetize the periosteum if possible. Perform local infiltration of subcutaneous tissues in both medial and cephalad directions to achieve adequate anesthesia of tissues at the intended path of the Tuohy needle and epidural catheter. Introduce the epidural needle with the bevel directed cephalad perpendicular to the anesthetized skin and advance until the ipsilateral lamina or transverse process is contacted. If lamina is not contacted, care may be taken to avoid advancing the needle laterally, which will place the needle in the paravertebral space. The needle depth to the lamina is then noted, and the needle is withdrawn back to skin and advanced again slightly medially; this step is repeated until the needle contacts bone at a slightly more superficial (approximately 2-5 mm) depth than the original depth at the lateral lamina. This suggests the epidural needle tip is midline at the junction of the lamina and spinous process (not shown). The needle is withdrawn and advanced with the same medial angle but in small increments cephalad to the same depth. Either bone or ligamentum flavum is contacted. If bone is contacted, the needle is redirected cephalad and advanced. If bone is no longer contacted and the depth exceeds the depth previously noted, the epidural needle stilette is removed. The luer lock loss-of-resistance syringe is attached to the needle for loss of resistance. Once loss of resistance is attained, stabilize the epidural needle and thread the catheter. Secure the catheter using a sterile locking device and adherent dressings. (1)induction of General anesthesia using 1Mg/kg fentanyl then propofol 2mg/kg and roucronioum 0.5mg/kg then endotracheal tube (ETT) insertion in the trachea via glottis opening then starting mechanical ventilation with tidal volume (Tv) 7cm/kg, respiratory rate RR12, PEEP 7 and both TV&RR can be changed up and down to adjust EtCo2 in the range (30-35)mmHg ,then roucuronum dosing of 0.2 of the original full bolus dose every 40 minutes and Inhalational anesthesia of Isoflurane 1MAC any incident of postoperative, Hypotension ( mean arterial blood pressure (MBP) less than 60 mmHg, will be managed by using ephedrine bolus doses of 6mg , 300ml colloid voluven and in case if sever bleeding >20% Blood volume loss blood and plasma transfusion according to patients requirements. Bradycardia (HR less than 60 b/m.) will be managed by atropine bolus of 0.5 mg. Desaturation (SaO2< 90%) will be managed by increase oxygen ventilation fraction and bilateral chest auscultation for chest wheezing and increased air way pressure to exclude bronchospasm at the end of operation reversal drugs to be given after attaining the recovery criteria and extubation to be done in a smooth safe non stressful situation. Pain during the study postoperative period the 1st 24 hours after recovery will be managed using IV pethidine 0.5mg/kg blouse without using NSAIDs.
* Postoperative management: Monitoring NIBP, Puls, puls oximetry, ECG in the recovery room to complete 6 hours from the operation start time in the recovery room then sending the patient to the word .Pain will be assessed by VAS between 0 and 100 (0 representing no pain and 100 is the worst pain) postoperatively at 1,2, 6 hours. Total requirements of postoperative 1st 24 pethidine rescue analgesic requirement will be recorded Standing Orders for Epidural Combined Opioids and Local Anesthetic Infusions (nursing instructions) Keep IV access, don't remove. Hourly RR, sedation score, VAS, Dose administration 4hourly BLP HR, Temp. Priapism if occur requires immediate treatment 1st to stop epidural infusion. (A case is reported of a 45-year-old male patient in which a clear relation is demonstrated between continuous thoracic epidural analgesia and priapism after transabdominal nephrectomy.) (9)

Call on-call anesthesia doctor if, RR<8, VAS>3, sedation score ≥3, systolic BP <100 mmHg, HR<50 B/minute Stop infusion if RR<8/min or sedation score=3-4, and if Priapism occur. Management …naloxone 0.1 mg IV bolus repeat every 5minutes till RR >10 and patient becomes responsive

ELIGIBILITY:
Inclusion Criteria:

1. Nephrectomy surgery
2. ASA I-III
3. Both sexes
4. Age 18 - 65 years. -

Exclusion Criteria:

1-Patient refusal of epidural cathetar insrtion 2-Morbid obesity BMI>35 3- Hypersensitivity to amide local anesthetics, opioid fentanyl. 4-Contraindications to epidural anesthesia (coagulopathies), 5-Cardiac disease, hepatic disease, renal or respiratory failure, and Diseased both kidneys.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
postoperative pain using 100mm VAS | 6 hours of epidural infusion stopped compared to basal (just on stopping the infusion
  postoperative pain during rest (lying supine), deep inspiration, coughing, and movement (getting up from supine to sitting position) using 100mm VAS

SECONDARY OUTCOMES:
postoperative IV rescue analgesic | total dose in the postoperative 1st 24hours
  postoperative analgesic request total dose
Mean arterial blood pressure | intraoperative every 1hour and every 2 hours for 1st postoperative 6 hours
  intraoperative & postoperative
Heart rate | intraoperative every 1hour and every 2 hours for 1st postoperative 6 hours
  intraoperative & postoperative
puls oxymeter desaturation | intraoperative every 1hour and every 2 hours for 1st postoperative 6 hours
  intraoperative & postoperative
Ramsy sedation score | basal and every 2 hours for the next 6 postoperative hours after recovery
  sedation scoreIf Awake Ramsey 1=Anxious, agitated, restless Ramsey 2=Cooperative, oriented, tranquil Ramsey 3=Responsive to commands only Ramsey 4=Brisk response to light glabellar tap or loud auditory stimulus Ramsey 5=Sluggish response to light glabellar tap or loud auditory stimulus Ramsey 6=No response to light glabellar tap or loud auditory stimulus
Modified Bromage score | basal every 2 hours for the next 6 postoperative hours after recovery
  1
  Complete block (unable to move feet or knees)
  2
  Almost complete block (able to move feet only)
  3
  Partial block (just able to move knees)
  4
  Detectable weakness of hip flexion while supine (full flexion of knees)
  5
  No detectable weakness of hip flexion while supine
  6
  Able to perform partial knee bend
Postoperative itching | incidence during 1st 24 hours after surgery.
  incidence yes or no
Postoperative Vomiting | incidence during 1st 24 hours after surgery.
  incidence yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. ghanem, A.professor, Principal Investigator — associate Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura Urology and Nephrology Center-Mansoura Univeristy, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided